CLINICAL TRIAL: NCT04003831
Title: Navigated Peripheral OCT Imaging With the P200TxE
Brief Title: Navigated OCT Imaging With the P200TxE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OPT1033
Record Dates: First submitted 2019-06-12; First posted 2019-07-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Optical Coherence Tomographer (Other)
  Interventions: Device: Device: P200TxE

INTERVENTIONS:
Device: Device: P200TxE — The P200TxE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.

SUMMARY:
The P200TxE will be used to obtain peripheral OCT (optical coherence tomography) images.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site,
3. Subjects who agree to participate in the study;
4. Subjects presenting with some form of peripheral retina pathology or retina pathology with peripheral manifestations.

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Qualitative Assessment of OCT Clinical Utility | 1 year
  Clinical utility of the OCT scans will be assessed from the clinician questionnaire using a four point scale.
Qualitative Assessment of OCT Scan Quality | 1 year
  Image quality of the OCT scans will be assessed from the clinician questionnaire using a four point scale.

SECONDARY OUTCOMES:
Safety Assessment from Adverse Events | 1 year
  Analysis of safety will be assessed through adverse events reported by the site and documented on each subject's case report form.

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Consultants of San Diego, Poway, California, United States

IPD SHARING:
Plan to Share IPD: No